CLINICAL TRIAL: NCT00438984
Title: Phase I Study To Evaluate Cellular Adoptive Immunotherapy Using Autologous CD8+ Antigen-Specific T Cell Clones Following Cyclophosphamide Conditioning For Patients With Metastatic Melanoma
Brief Title: Therapeutic Autologous Lymphocytes, Cyclophosphamide, and Aldesleukin in Treating Patients With Stage IV Melanoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Yee, Cassian, Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Organization: Fred Hutchinson Cancer Center (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2140.00; NCI-2010-01280 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); R21CA128283 (NIH)
Record Dates: First submitted 2007-02-20; First posted 2007-02-22 (Estimated); Last update posted 2012-03-16 (Estimated); Status verified 2012-03

CONDITIONS: Recurrent Melanoma; Stage IV Melanoma
MeSH Terms: conditions — Melanoma | interventions — Cyclophosphamide; aldesleukin; Interleukin-2; Immunohistochemistry; Biopsy; Immunologic Techniques; Polymerase Chain Reaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (chemotherapy, immunosuppressive, lymphocytes) (Experimental): All patients receive high-dose cyclophosphamide IV on days -3 and -2 and autologous antigen-specific cytotoxic CD8+ T-lymphocyte clones IV over 30-60 minutes on day 0.
  COHORT I: Beginning within 6 hours of T cell infusion, patients receive low-dose aldesleukin SC twice daily on days 0-14.
  COHORT II: Beginning within 6 hours of T cell infusion, patients receive high-dose aldesleukin IV 3 times daily on days 0-5.
  Interventions: Drug: cyclophosphamide; Biological: therapeutic autologous lymphocytes; Biological: aldesleukin; Other: immunohistochemistry staining method; Procedure: biopsy; Other: laboratory biomarker analysis; Other: immunologic technique; Genetic: polymerase chain reaction

INTERVENTIONS:
Drug: cyclophosphamide — Given IV
  Other Names: CPM; CTX; Cytoxan; Endoxan; Endoxana
Biological: therapeutic autologous lymphocytes — Given IV
  Other Names: AL; Autologous Lymphocytes; autologous T cells
Biological: aldesleukin — Given IV or SC
  Other Names: IL-2; Proleukin; recombinant human interleukin-2; recombinant interleukin-2
Other: immunohistochemistry staining method — Correlative studies
  Other Names: immunohistochemistry
Procedure: biopsy — Optional correlative studies
  Other Names: biopsies
Other: laboratory biomarker analysis — Correlative studies
Other: immunologic technique — Correlative studies
  Other Names: immunological laboratory methods; laboratory methods, immunological
Genetic: polymerase chain reaction — Correlative studies
  Other Names: PCR

SUMMARY:
RATIONALE: Biological therapies, such as therapeutic autologous lymphocytes, may stimulate the immune system in different ways and stop tumor cells from growing. Drugs used in chemotherapy, such as cyclophosphamide, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Cyclophosphamide may also stimulate the immune system in different ways and stop tumor cells from growing. Aldesleukin may stimulate white blood cells to kill tumor cells. Giving therapeutic autologous lymphocytes together with cyclophosphamide and aldesleukin may be an effective treatment for melanoma.

PURPOSE: This phase I trial is studying the side effects of giving therapeutic autologous lymphocytes together with cyclophosphamide and aldesleukin in treating patients with stage IV melanoma

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the safety and toxicity of cellular adoptive immunotherapy in melanoma patients receiving autologous CD8+ antigen-specific T cell clones following cyclophosphamide conditioning and post-infusion IL-2.

II. To assess the duration of in vivo persistence of adoptively transferred CD8+ T cell clones.

SECONDARY OBJECTIVES:

I. Evaluate the antitumor effect of adoptively transferred CD8+ antigenspecific cytotoxic t lymphocytes (CTL) clones following cyclophosphamide conditioning and post-infusion IL-2.

OUTLINE:

Patients are assigned 1of 2 treatment cohorts.

All patients receive high-dose cyclophosphamide intravenously (IV) on days -3 and -2 and autologous antigen-specific cytotoxic CD8+ T lymphocyte clones IV over 30-60 minutes on day 0.

COHORT I: Beginning within 6 hours of T cell infusion, patients receive low-dose aldesleukin subcutaneously (SC) twice daily on days 0-14.

COHORT II: Beginning within 6 hours of T cell infusion, patients receive high-dose aldesleukin IV 3 times daily on days 0-5.

Treatment continues in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 4 weeks, 8 weeks, and every 3 months thereafter for up to 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Histopathological documentation of melanoma concurrent with the diagnosis of metastatic disease
* Expression of HLA-A2, B44, or A3 as determined by Fred Hutchinson Cancer Research Center (FHCRC) human leukocyte antigen (HLA) typing lab
* Zubrod performance status of 0-1
* Bi-dimensionally measurable disease by palpation on clinical exam, or radiographic imaging (X-ray, CT scan)
* Normal cardiac stress test within 182 days prior to enrollment is required of all patients over 50 years old or those with an abnormal electrocardiogram (ECG), any history of cardiac disease, a family history of cardiac disease, hypercholesterolemia or hypertension
* FOR LEUKAPHERESIS:
* Pulse > 45 or < 120
* Weight >= 45 kg
* White blood cell count (WBC) >= 3,000
* Temperature =< 38C (=< 100.4 F)
* Hematocrit (HCT) >= 30%
* Platelets >= 100,000
* FOR T CELL INFUSION: Patients must be willing and able to discontinue the use of all anti-hypertensive medications 24 hours prior to and during IL-2 therapy

Exclusion Criteria:

* Pregnant women, nursing mothers, men or women of reproductive ability who are unwilling to use effective contraception or abstinence; women of childbearing potential must have a negative pregnancy test within two weeks prior to entry
* Serum creatinine > 1.6 mg/dL or Creatinine clearance < 75 ml/min
* Serum glutamic oxaloacetic transaminase (SGOT) > 150 IU or > 3x upper limit of normal
* Bilirubin > 1.6 mg/dL
* Prothrombin time > 1.5 x control
* Clinically significant pulmonary dysfunction, as determined by medical history and physical exam; patients so identified will undergo pulmonary functions testing and those with forced expiratory volume in one second (FEV1) < 2.0 L or carbon monoxide diffusing capacity (DLco) (corr for Hgb) < 75% will be excluded
* Significant cardiovascular abnormalities as defined by any one of the following:
* Congestive heart failure;
* Clinically significant hypotension;
* Symptoms of coronary artery disease;
* Presence of cardiac arrhythmias on electrocardiograph (EKG) requiring drug therapy;
* Ejection fraction < 50 % (echocardiogram or multi gated acquisition scan [MUGA])
* Symptomatic central nervous system metastases greater than 1 cm at the time of therapy; patients with 1-2 asymptomatic, less than 1 cm brain/central nervous system (CNS) metastases without significant edema may be considered for treatment; if sub-centimeter CNS lesions are noted at study entry, than a repeat imaging will be performed if more than 3 weeks have elapsed from the last scan; patients will not be treated if CNS lesions are > 1 cm or if patient is symptomatic from brain metastasis
* Patients with active infections or oral temperature > 38.2 C within 72 hours of study entry or systemic infection requiring chronic maintenance or suppressive therapy
* Chemotherapeutic agents (standard or experimental), radiation therapy, or other immunosuppressive therapies less than 3 weeks prior to T cell therapy; (patients with bulky disease may undergo cytoreductive chemotherapy but treatment will be discontinued at least 3 weeks prior to T cell therapy)
* Clinically significant autoimmune disorders or conditions of immunosuppression; patients with acquired immune deficiency syndrome (AIDS) or human immunodeficiency virus (HIV)-1 associated complex or known to HIV antibody seropositive or known to be recently polymerase chain reaction (PCR)+ for hepatitis are not eligible for this study; virology testing will be done within 6 months of T cell infusion; the severely depressed immune system found in these infected patients and the possibility of premature death would compromise study objectives
* FOR T CELL INFUSION: Patients with active infections or oral temperature > 38.2 C within 72 hours of study entry or systemic infection requiring chronic maintenance or suppressive therapy
* FOR T CELL INFUSION: Chemotherapeutic agents (standard or experimental), radiation therapy, or other immunosuppressive therapies less than 3 weeks prior to T cell therapy
* FOR T CELL INFUSION: Current treatment with steroids
* FOR T CELL INFUSION: Patients must not be receiving any other experimental drugs within 3 weeks of the initiation of the protocol and must have recovered from all side effects of such therapy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2006-12; Primary Completion 2011-01 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
The identification of a CY/IL-2 regimen that is considered to be safe | Baseline, 4 weeks and 8 weeks
The identification of a CY/IL-2 regimen (among those considered safe) which yields the greatest effect on the duration of in vivo persistence of adoptively transferred CTL clones | Baseline, 4 weeks and 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Cassian Yee, Principal Investigator — Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Locations (1):
- Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington, United States